CLINICAL TRIAL: NCT03585790
Title: The Impact of Soft Contact Lens Attributes on Symptoms Associated With Digital Eye Strain in Symptomatic Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pete Kollbaum, OD, PhD (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Pete Kollbaum, OD, PhD, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Kollbaum001
Record Dates: First submitted 2018-04-26; First posted 2018-07-13 (Actual); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Asthenopia; Myopia
Keywords: Eye Fatigue
MeSH Terms: conditions — Asthenopia; Myopia | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multifocal Optics first, then Single Vision Optics (Other): First Intervention (1 week) Second Intervention (1 week)
  Interventions: Device: Contact lens with Multifocal Optics; Device: Contact lens with Single Vision Optics
- Single Vision Optics first, then Multifocal Optics (Other): First Intervention (1 week) Second Intervention (1 week)
  Interventions: Device: Contact lens with Multifocal Optics; Device: Contact lens with Single Vision Optics

INTERVENTIONS:
Device: Contact lens with Multifocal Optics — This contact lens has optics to aid the accommodative and convergence systems
Device: Contact lens with Single Vision Optics — This contact lens has standard single vision optics

SUMMARY:
Despite its prevalence, the ocular causes of eye fatigue or unknown and may be related to the cornea/contact lens surface, the accommodative system, the convergence system, overall postural/muscle fatigue, or a combination of these or other causes. The current study aims to systematically investigate the incremental benefits in ameliorating eye fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported "eye fatigue" at least once per week attributable to digital device use with baseline.
2. Uses a digital device (phone, tablet, computer, etc) at least 4 hours per day
3. Mobile digital device with active data and text plan, able to receive email and text messages
4. Habitual 2-week or monthly silicone single vision hydrogel soft contact lens use; habitually wearing lenses for 6 or more hours per day for 5 or more days per week for the past 30 days
5. Habitual soft contact lens prescription optimized over-refraction within ±0.25 D
6. 18-35 years of age
7. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
8. Vertex corrected refractive cylinder must be -0.75 or less.
9. Visual acuity best correctable to 20/25 or better for each eye
10. The subject must read and sign the Informed Consent form.

Exclusion Criteria:

1. A habitual wearer of any of the test lenses
2. Any active conditions that may prevent soft contact lens wear.
3. Any doctor diagnosed, self-reported ocular surface disease or dry eye requiring regular, ongoing treatment
4. Any doctor diagnosed, self-reported accommodative or binocular vision issues
5. History of issues of eye alignment or binocularity by self-report

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Clinical Optics Research Lab, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (1 Week)
Arm/Group | Multifocal Optics First, Then Single Vision Optics | Single Vision Optics First, Then Multifocal Optics
Started (First intervention) | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Multifocal Optics First, Then Single Vision Optics | Single Vision Optics First, Then Multifocal Optics
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifocal Optics First, Then Single Vision Optics | Single Vision Optics First, Then Multifocal Optics | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.87 (3.37) | 22.5 (3.01) | 22.17 (3.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 16 | 37
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Eye Fatigue
Description: Subjective Rating of Eye Fatigue, response to question "How would you rate your overall eye fatigue/tiredness?" on a 0-100 slider visual analog scale, where 0 represents 'Not Noticeable' and 100 represents 'Very Noticeable', with the numerical representation of their visual analog selection displayed to the right of the slider scale. Score reported is rating as described above.
Time Frame: 1 week
Population: Outcome measures reported for both groups combined secondary to crossover design.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Multifocal Optics First, Then Single Vision Optics | Single Vision Optics First, Then Multifocal Optics | Total
Number analyzed (Participants) | 23 | 22 | 45
units on a scale
  Single Vision | 18 [6.5 to 39] | 21 [15.25 to 48] | 21 [11 to 45]
  Multifocal | 17 [6.5 to 33.5] | 21.5 [16.75 to 38.75] | 20 [8 to 38]
Statistical Analysis 1: Comparison: Multifocal Optics First, Then Single Vision Optics; Ho: Single Vision - Multifocal >= M vs. Ho: Single Vision - Multifocal < M. Alpha = 0.05, two sided beta = 0.80; Test type: Non-Inferiority — Margin acceptable mean difference (Single Vision - Multifocal) = -5 rating units (0-100 scale, 0 = optimal); p = 0.18, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 month
Arm/Group | Multifocal Optics First, Then Single Vision Optics | Single Vision Optics First, Then Multifocal Optics
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03585790/Prot_SAP_000.pdf